CLINICAL TRIAL: NCT04392856
Title: Transdiagnostic Treatment of Emotional Disorders for Women in a Homeless Situation
Acronym: UPHW
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); University of Alcala (Other); Council of Madrid (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEM2016-75317-R
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2020-05

CONDITIONS: Anxiety; Depression
Keywords: Unified Protocol; Transdiagnostic approach; Homelessness
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: All women in a homeless situation attending any of the collaborating shelters will be asked to participate in the present study. Once inclusion criteria are met, each participant will be assigned to experimental condition or control condition.
  This research is composed by two sequential studies. The first study will deliver the UP in a group format, while the second study will deliver the UP on a one-to-one basis. Since these studies will not be performed concurrently, women will be assigned within each study to intervention or control condition. In the first study, participants will be assigned to one of two conditions: experimental condition (Unified Protocol, UP in group delivery) or waitlist control condition (WLC). In the second study, participants will be assigned to one of two conditions: experimental condition (Unified Protocol, UP in individual delivery) or control condition (WLC).
Who Masked: Outcomes Assessor
Masking Description: Participants will know if they are assigned to the treatment condition or to the WLC group. Shelter professionals and researchers will know the condition of each participant, however, independent evaluators will not know whether the woman is in UP or Waitlist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol Transdiagnostic Treatment Emotional Disorders (Experimental): An adaptation of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) to women in a homeless situation will be implemented in public shelters setting in Madrid, Spain.
  The UP adaptation is an intervention based protocol for emotional disorders, consisted of 12 treatment sessions of one and a half hours of duration each, at a rate of one per week.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP)
- Waitlist Control condition (Other): The participants assigned to the waitlist control condition will not immediately receive the intervention. They will wait for 3 months, which is the duration of the intervention in the experimental group. After that time, they will be offered the same psychological treatment as those assigned to the UP (experimental condition).
  Interventions: Behavioral: Same than experimental condition (UP), after it finishes

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP) — The Spanish Version of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders for Homeless Women. The protocol contains five modules: (1) mindful emotion awareness, (2) cognitive flexibility, (3) countering emotional behaviors, (4) recognizing and confronting physical sensations, and (5) emotion exposures. This adaptation of Unified Protocol is organized in twelve sessions: Emotional disorders and emotional regulation; Motivation for change; Understanding the role of emotions; Mindful emotion awareness, Cognitive flexibility, Understanding and confronting physical sensations, Countering emotional behaviors, Emotional avoidance, Emotion exposure; Achievement recognition and look to the future; and Relapse prevention and closure.
  Arms: Unified Protocol Transdiagnostic Treatment Emotional Disorders
Behavioral: Same than experimental condition (UP), after it finishes — The Spanish Version of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders for Homeless Women. The protocol contains five modules: (1) mindful emotion awareness, (2) cognitive flexibility, (3) countering emotional behaviors, (4) recognizing and confronting physical sensations, and (5) emotion exposures. This adaptation of Unified Protocol is organized in twelve sessions: Emotional disorders and emotional regulation; Motivation for change; Understanding the role of emotions; Mindful emotion awareness, Cognitive flexibility, Understanding and confronting physical sensations, Countering emotional behaviors, Emotional avoidance, Emotion exposure; Achievement recognition and look to the future; and Relapse prevention and closure.
  Arms: Waitlist Control condition

SUMMARY:
The aim of this study is to assess the effectiveness and feasibility of an adaptation of the Unified Protocol (UP) for Transdiagnostic Treatment of Emotional Disorders to women living homeless in Madrid, Spain. To address this goal, both clinical and psychosocial outcomes will be measured. The application of the UP is postulated as an effective tool for improving mental health and well-being of women in a homeless situation, which in turn will enhance their social inclusion process.

DETAILED DESCRIPTION:
The European Strategy for the Homeless People states that homelessness is the most extreme form of poverty and exclusion, which violates human dignity and poses a risk to health and life. Women constitute a particularly vulnerable subgroup among homeless people. Women living homeless show significant deterioration in their psychological welfare and mental health, which, among other aspects, is an obstacle in the access to care resources and inclusion processes.

There is a growing interest in the effectiveness and efficiency of intervention techniques to address mental health problems. The high comorbidity between mental health disorders, and especially emotional disorders, has promoted the development and consolidation of a transdiagnostic perspective. This perspective raises the existence of common mechanisms involved in the maintenance of different disorders, so that there would be a preamble to cognitive and/or behavioral processes shared by various psychological disorders. The design of a transdiagnostic treatment strategy allows a more inclusive approach to mental health and facilitates the design of similar treatment programs applicable to a wide range of mental disorders. Therefore, the transdiagnostic treatment could be a feasible and effective alternative to address some of the most common problems in mental health among women in a homeless situation. This approach could be useful to improve a diversity of symptoms in the own context of homeless living women and facilitate a systematic evaluation of its effectiveness.

The overall objective of this project is the development of a feasible and effective intervention adapted to the needs of women in a homeless situation and the service resources where they are attended. Moreover, the project aims to compare the group versus individual delivery of the UP among women in a homeless situation. This research is based on the hypothesis that the UP adaptation, both in group and individual delivery, will be effective in reducing anxiety and depression symptoms, decreasing negative affect and increasing psychological well-being, health state, positive affect, social support and quality of life. Strengths but also barriers and difficulties encountered in each format of intervention will be examined. This knowledge will be key to develop specific and adapted materials that enable effective interventions practices in the services resources for homeless people.

The UP intervention will consist of 12 weekly sessions lasting an hour and a half, applied in different centers for homeless people in Madrid. There will be several assessment moments: before the intervention, twelve intersession assessments (i.e., one per session), after the intervention, and 3 months, 6 months and 9 months follow-ups. The psychological intervention will be carried out by therapists with a background in psychology.

With this research it is expected to achieve results with impact at the technical level (in the design of effective interventions for psychological treatment of women in a homeless situation), on a scientific level (expanding knowledge about the effectiveness of intervention programs for women in social exclusion situations), and, especially, at the social level (affecting the quality of life and the processes of social inclusion of women in a homeless situation).

ELIGIBILITY:
Inclusion Criteria:

* Being a woman.
* Being aged over 18 years old.
* Providing written, informed consent.
* The participant is fluent in the language in which the treatment and evaluation are performed (i.e. Spanish).
* Being able to attend to the evaluation and treatment sessions
* Having access to the shelters where the intervention will be carried out.

Exclusion Criteria:

* Being diagnosed with a severe mental disorder in active phase (i.e. schizophrenia, bipolar disorder or an organic mental disorder).
* Being diagnosed a severe cognitive deterioration.
* Being under alcohol or substance effects when the pre-assessment is carried out.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Change in the Beck Depression Inventory (BDI-II) (Beck, Steer, & Brown, 1990); Spanish adaptation (Sanz, Navarro, & Vázquez, 2003) at pre, post intervention and at 3, 6 and 9 month follow-ups. | Up to 9 months
  The BDI-II is a 21-item self-report measure designed to assess depression severity. Each item is rated from 0 to 3 with a total score of a maximum of 63 points. The Spanish version has shown good internal consistency (α = 0.86).
Change in the Beck Anxiety Inventory (BAI) (Beck, & Steer, 1993); Spanish adaptation (Magán, Sanz, & García-Vera, 2008) at pre, post intervention and at 3, 6 and 9 month follow-ups. | Up to 9 months
  The BAI is a 21-item self-report measure designed to assess anxiety severity. Each item has a 4-point severity scale (e.g., not at all, mildly, moderately, and severely), addressing symptoms experienced during the past week. The internal consistency of the Spanish version has been found to range from .85 to .94.

SECONDARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS) (Watson, Clarck, & Tellegen, 1988); Spanish adaptation (López-Gómez, Hervás, & Vázquez, 2015) at pre, post intervention and at 3, 6 and 9 month follow-ups | Up to 9 months
  The PANAS is a 20-item self-report measure designed to assess negative and positive affect in the last week. Each item has a 5-point severity scale (e.g., not at all, mildly, moderately, quite a lot, and severely) with a total score from 20 to 100. The internal consistency of the Spanish version was .92 for positive affect subscale and .88 for negative affect subscale.
Change in the Pemberton Happiness Index (PHI) (Hervás & Vázquez, 2013) at pre, post intervention and at 3, 6 and 9 month follow-ups | Up to 9 months
  The PHI is a 21-item measure designed to assess integrative well-being using a scale from 0 (fully disagree) to 10 (fully agree) in the first 11 items and dichotomy answers (yes/no) in the last 10 items. It includes two subscales: remember well-being (general, hedonic, eudaimonic, and social well-being) and experienced well-being. Cronbach´s alpha of Spanish version was .84.
Change in the Short-Form Health Survey Health Questionnaire (SF-12) (Ware, Kosinski, & Keller, 1996); Spanish adaptation (Vilagut et al., 2008) at pre, post intervention and at 3, 6 and 9 month follow-ups | Up to 9 months
  The SF-12 is a generic health status instrument with 12 items, and eight subscales (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health). These eight subscales can be combined into two scores for physical health (PH) and mental health (MH), and a total score, ranged from 0 to 100, where higher scores reflect better self-reported health. The internal consistency of the Spanish version was α = .85 for PH and α = .78 for MH.
Change in the Social Support Questionnaire (SSQ) (Sarason, Sarason, Shearin, & Pierce, 1987); Spanish adaptation (Martínez-López et al., 2014) at pre, post intervention and at 3, 6 and 9 month follow-ups. | Up to 9 months
  The SSQ is a 6 items measure of social support. It includes two scales: number and satisfaction with social support (on a scale ranging from 1 to 9). The Spanish version has shown good internal consistency for both dimensions (α = 0.90 and α = 0.93, respectively).
Change in the Satisfaction with Life Domain Scale (SLDS) (Baker e Intagliatta, 1982); Spanish version by Muñoz, Panadero, & Rodríguez (2010) at pre, post intervention and at 3, 6 and 9 month follow-ups. | Up to 9 months
  This questionnaire was adapted for use in rehabilitation centers for people with mental disorders by Muñoz et al. (2010). It is a 18-item self-report measure that was designed for assessing their actual satisfaction in various aspects of the life. An 8-point visual analog scale with faces is used.
Overall Depression Severity and Impairment Scale (ODSIS) (Bentley, Gallagher, Carl, Barlow, 2014); Spanish version (Mira et al., 2019) at intersession assessment | Up to 3 months
  The ODSIS is a 5-item self-report measure that was designed for assessing the frequency and intensity of depression symptoms, the functional impairment related to these depressive symptoms, as well as behavioral avoidance across emotional disorders over the past week. Response items are coded from 0 to 4 and can be summed to obtain a total score ranging from 0 to 20. The internal consistency of the Spanish version was between .91 and .94.
Overall Anxiety Severity and Impairment Scale (OASIS) (Norman, Cissell, Means-Christensen, & Stein, 2006); Spanish version (González-Robles et al., 2018) at intersession assessment | Up to 3 months
  The OASIS is a self-report questionnaire designed to evaluate the severity and functional impairment associated with anxiety. The scale presents five items with a 5-point likert scale ranging from 0 (I didn't feel anxious) to 4 (Constant anxiety). The total scale score, which ranges from 0 to 20, is obtained by summing all items. Cronbach's alpha of the Spanish version was 0.86.

OTHER OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) (Saunders et al. 1993); Spanish adaptation (Rubio, Bermejo, Caballero, & Santo Domingo, 1998). | Up to 9 months
  The AUDIT was developed as a simple screening method for excessive alcohol consumption. The AUDIT consists of 10 questions about the level of consumption, symptoms of dependence and alcohol-related consequences with a total score of a maximum of 63 points. The Spanish version reliability coefficient was 0.86.
Drug Abuse Screening Test (DAST-10) (Skinner, 1982); Spanish adaptation (Pérez-Gálvez et al., 2010) | Up to 9 months
  It is one of the instruments more used for detection is the Drug Abuse Screening Test (DAST). The DAST-10 is a 10 items self-reports with dichotomous response (yes/no). The Spanish version has shown a high internal consistency (α = 0.89).

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Panadero, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Faculty of Psychology. Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marin C, Guillen AI, Rodriguez-Moreno S, Dieguez S, Panadero S, Farchione T. Application of the unified protocol for transdiagnostic treatment of emotional disorders among homeless women: A feasibility study. Psychotherapy (Chic). 2021 Jun;58(2):242-247. doi: 10.1037/pst0000357. Epub 2021 Feb 4. PMID 33539144